CLINICAL TRIAL: NCT01083290
Title: Pharmacokinetic Study of Spironolactone 25 mg, 50 mg and 100 mg Tablets in Healthy Subjects Under Fasting Conditions.
Brief Title: Pharmacokinetic Study of Spironolactone 25 mg, 50 mg and 100 mg Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Ulla Sairanen/ Clinical Study Manager, Orion Corporation Orion Pharma
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 0300012
Record Dates: First submitted 2010-03-08; First posted 2010-03-09 (Estimated); Last update posted 2010-05-10 (Estimated); Status verified 2010-05

CONDITIONS: Healthy
Keywords: spironolactone; linearity of pharmacokinetics; Healthy volunteers
MeSH Terms: interventions — Spironolactone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Order of strenghts; 25 mg, 50 mg, 100 mg (Experimental)
  Interventions: Drug: Spironolactone
- Order of strenghts; 50 mg, 100 mg, 25 mg (Experimental)
  Interventions: Drug: Spironolactone
- Order of strenghts; 100 mg, 25 mg, 50 mg (Experimental)
  Interventions: Drug: Spironolactone

INTERVENTIONS:
Drug: Spironolactone — single dose of one tablet; 25 mg tablet
Drug: Spironolactone — single dose of one tablet; 50 mg tablet
Drug: Spironolactone — single dose of one tablet; 100 mg tablet

SUMMARY:
Objective is to investigate pharmacokinetics and to estimate the level of dose linearity of spironolactone and its metabolites canrenone and 7α-thiomethylspirolactone from Spironolactone 25 mg, 50 mg and 100 mg Tablets

ELIGIBILITY:
Inclusion Criteria:

* Subjects with normal findings as determined by baseline history, physical examination and vital signs, haemogram, biochemistry, infectious disease screening, urinalysis, 12 lead ECG

Exclusion Criteria:

* Any condition requiring regular concomitant medication or likely to need any concomitant medication during the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2010-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Cmax, AUC0-t and AUC0-inf of Spironolactone and its metabolites canrenone and 7α-thiomethylspirolactone in plasma | up to 72 h after the study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Suhas Khandave, MD, Principal Investigator — Accutest Research Laboratories (I) Pvt. Ltd.
Locations (1):
- Accutest Research Laboratories (I) Pvt. Ltd., Mumbai, India